CLINICAL TRIAL: NCT01415583
Title: Evaluating Perioperative Dexamethasone and the Risk of Bleeding in Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Christopher Hartnick, M.D., Director, Division of Pediatric Otolaryngology, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-03-016
Record Dates: First submitted 2010-10-27; First posted 2011-08-12 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Post-operative Hemorrhage
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): Placebo is described in chart
  Interventions: Drug: Dexamethasone
- Dexamethasone (Experimental): Dexamethasone is described in chart
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — 0.5mg/kg (max dose 20mg)
  Other Names: Decadron

SUMMARY:
Tonsillectomy (removal of the tonsils) is a very common surgery in children. Bleeding after tonsillectomy is one of the risks of this surgery and can be more dangerous in children since they have less blood volume than adults. In order to improve recovery after tonsillectomy, steroids (medication that is a strong anti-inflammatory) are often given during the surgery. Recently, a study showed steroids given at the time of tonsillectomy increase the risk of bleeding significantly over children who did not receive steroids. This finding has raised concerns in the Ear, Nose, and Throat (ENT) community since most ENT's use steroids during tonsillectomy in children. The investigators look to explore this question further.

To answer the question of whether perioperative steroid administration significantly affects the rate of post-tonsillectomy bleeding, the investigators propose to test the following hypotheses in a prospective, randomized, blinded placebo-controlled trial: dexamethasone does not cause an increase in post-operative bleeding rate in tonsillectomy.

DETAILED DESCRIPTION:
Detailed description is entered above

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 3 to 18 undergoing tonsillectomy or adenotonsillectomy by electrocautery alone for the indication of sleep disordered breathing or infectious tonsillitis.
* Patients with complex medical conditions or craniofacial abnormalities will be included.
* Informed consent and child assent are required for enrollment.
* Eligibility will be determined by the principal investigator, associate investigator or research nurse.

Exclusion Criteria:

* Subjects with a known personal or family history of any bleeding disorder will be excluded.
* Subjects currently on oral corticosteroids for other medical conditions or have recently taken any oral corticosteroid within two weeks of surgery.
* Patients with tonsillectomy performed using a cold knife technique, microdebrider, coblation or plasma knife due to surgeon or parent preference.
* Where appropriate subjects who do not have informed consent or child assent signed will be excluded
* Children less than three years old will be excluded due to the fact the majority of these children at the collaborating centers have an adenotonsillectomy using the microdebrider for pain control purposes.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 314 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hartnick, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gallagher TQ, Hill C, Ojha S, Ference E, Keamy DG, Williams M, Hansen M, Maurer R, Collins C, Setlur J, Capra GG, Brigger MT, Hartnick CJ. Perioperative dexamethasone administration and risk of bleeding following tonsillectomy in children: a randomized controlled trial. JAMA. 2012 Sep 26;308(12):1221-6. doi: 10.1001/2012.jama.11575. PMID 23011712

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline | Dexamethasone
Started | 157 | 157
Completed | 157 | 157
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Dexamethasone | Total
Number analyzed (Participants) | 157 | 157 | 314
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6 [4 to 9] | 6 [4 to 8] | 6 [4 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 75 | 144
  Male | 88 | 82 | 170

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-tonsillectomy Bleeding
Time Frame: 2 weeks after surgery
Measure: Number (97.5% Confidence Interval); unit: participants
Arm/Group | Saline | Dexamethasone
Number analyzed (Participants) | 157 | 157
participants | 13 [10.4 to 15.6] | 17 [14.4 to 19.6]
Statistical Analysis 1: Comparison: Saline vs Dexamethasone; Test type: Non-Inferiority — Consistent with the noninferiority design, the null hypothesis states that the bleeding rate in patients receiving perioperative dexamethasone differed from the bleeding rate in patients receiving perioperative placebo; the alternative hypothesis states that the bleeding rate with dexamethasone is not greater than placebo by more than the noninferiority margin; p = 0.05, t-test, 1 sided
Statistical Analysis 2: Comparison: Saline vs Dexamethasone; Test type: Non-Inferiority — This noninferiority margin was set at 5%, meaning a difference in bleeding rates that did not exceed 5% would be taken as evidence that the bleeding with dexamethasone is not greater than that with placebo by more than 5%; p = 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 6 months
Description: Subjects were instructed to inform study staff of any adverse events occurring during the 2 week post-operative period and during any follow-up visits 6 months post surgery.
Arm/Group | Saline | Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/157
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/157
Other Adverse Events (participants affected / at risk) | 0/157 | 0/157

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No